CLINICAL TRIAL: NCT05321329
Title: Adjuvant CAPECITABINE in High Risk PSEUDOMYXOMA PERITONEI Patients Treated With CYTOREDUCTIVE SURGERY (CRS) and HYPERTERMIC INTRAPERITONEAL CHEMOTHERAPY (HIPEC)
Brief Title: Adjuvant CAPECITABINE in High Risk PSEUDOMYXOMA PERITONEI Patients
Acronym: ACAPP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 36/18
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Pseudomyxoma Peritonei
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Open label, non-comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Capecitabine will be taken orally at dose of 1250 mg/m2 PO BID on days 1→14 every 3 weeks Cycles are to be repeated every 21 days for a total of 8 cycles
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is a deoxycytidine derivative and fluorouracil PRODRUG that is used as an ANTINEOPLASTIC ANTIMETABOLITE in the treatment of COLON CANCER; BREAST CANCER and GASTRIC CANCER.Capecitabine is a Nucleoside Metabolic Inhibitor. The mechanism of action of capecitabine is as a Nucleic Acid Synthesis Inhibitor.

SUMMARY:
This is a phase II, mono institutional, non comparative study, evaluating adjuvant capecitabine in patients affected by KRAS mutated Pseudomyxoma peritonei treated with cytoreductive surgery and HIPEC.

Patient will be treated with 8 cycles of the study regimen that include:

Capecitabine 1250 mg/m2 PO BID day 1-14 q21 days

DETAILED DESCRIPTION:
A previous phase II study evaluated the combination of systemic concurrent mitomycin C and capecitabine in advanced unresectable PMP.

Fifteen out of 39 patients benefited from chemotherapy in the form of either reductions in mucinous deposition or stabilisation of progressive pretreatment disease determined on CT scan. Notably, two patients, originally considered unresectable, underwent potentially curative cytoreductive surgery. One-year and two-year tumour-related survival rates for the 40 patients were 84% and 61%, respectively.

FOLFOX-4 chemotherapy was evaluated on 20 patients with unresectable or recurrent PMP, obtaining a 20% response rate and a 65% disease control rate, 2 patients originally considered unresectable underwent complete cytoreduction. Median PFS and median OS were 8 months and 26.2 months respectively.

In a retrospective review of MCP (mucinous cancer peritonei) patients who had undergone CRS/HIPEC with or without perioperative systemic chemotherapy (any regimen), postoperative chemotherapy was associated with longer PFS (13.6 months) compared to pre-operative treatment (6.8 months, P < 0.01) and CRS/HIPEC alone (7.0 months, P = 0.03).

The OS of patients treated with systemic chemotherapy after previous CRS and HIPEC appeared to be associated with the length of PFS after primary treatment (p=0.04).

KRAS and GNAS mutations were associated with worse progression-free survival (PFS) at univariate analysis (P = 0.006 and 0.011, respectively). At multivariate analysis, only KRAS mutations were independently associated with PFS (P = 0.012).

This is the rationale that induced us to carry out an evaluation and feasibility assessment of an adjuvant approach with oral capecitabine in patients affected by KRAS mutated PMP with extensive peritoneal disease, after cytoreductive surgery and HIPEC.

Twenty-eight cases (intention to treat) will be recruited in 3 years and followed-up for 2 years. Currently, the annual PMP case-volume submitted to CRS-HIPEC amounts approximately 25 in our center. Considering that approximately 65-70% of cases could present the KRAS mutated status, we will accrue 28 patients over the study period. With such a sample size, we estimate that the study power is of 76% in case of a 40% relative reduction in the hazard of PFS. We assumed an exponential distribution of event times, a baseline median PFS of 27 months, and the use of a one-sided test at the 10% significance level, a choice justified by the exploratory nature of the study.

Given the low level of evidence on the tolerance of Capecitabine alone in the systemic treatment of PMP, an independent safety board will perform a strict monitorization of the adverse events in the subset of first 10 recruited cases.

Twenty-eight cases (intention to treat) will be recruited in 3 years and followed-up for 2 years. Currently, the annual PMP case-volume submitted to CRS-HIPEC amounts approximately 25 in our center. Considering that approximately 65-70% of cases could present the KRAS mutated status, we will accrue 28 patients over the study period.[6] With such a sample size, we estimate that the study power is of 76% in case of a 40% relative reduction in the hazard of PFS. We assumed an exponential distribution of event times, a baseline median PFS of 27 months [6], and the use of a one-sided test at the 10% significance level, a choice justified by the exploratory nature of the study.

This study should be completed after 36 months enrolment, followed by 2 years of follow up. It is understood that these accrual rates are based on reasonable planning expectations.

Response to treatment has to be assessed after four cycles of treatment by using the same techniques used at baseline.(At baseline, each tumor lesions will be categorized in measurable or nonmeasurable; The measurable lesion can have longest diameter >20mm with conventional techniques (CT scan) or >10 mm with spiral CT scan;the non measurable lesions include the lesions with longest diameter <20 mm with conventional techniques (CT scan) or <10 mm with spiral CT scan and truly non measurable lesions;tumor lesion that are situated in a previously irradiated area might not be considered measurable).

Written informed consent must be obtained prior to the patients undergoing any study-specific procedures.Tumor assessment (TC/RMN abdomen plus TC thorax and PET) should be made within 28 days before treatment start.

Clinical assessment will be made up to 17 days before treatment start and includes: demographic data, medical history, electrocardiogram (ECG), CEA and Ca19.9 determination, pregnancy test, height, weight, vital signs (body temperature, blood pressure, pulse/heart rate), ECOG Performance Status, haematology, blood chemistry: bilirubin total and direct, AST/ALT, alkaline phosphatase, albumin, LDH, serum creatinine and estimated creatinine clearance (calculated using Cockcroft and Gault formula), glucose, electrolytes (sodium, potassium, calcium).

Study Medication: Capecitabine is available in the form of film-coated tablets in two strengths 150 mg and 500 mg. Capecitabine is to be administered orally twice daily within 30 minutes after the end of a meal (breakfast, dinner). Tablets should be swallowed with water (and not fruit juices). For capecitabine the investigator must calculate the body surface area (m2) of the patient. If there is a 10% decrease in body weight comparing to baseline, the BSA will be recalculated. If the calculated BSA is >2.2 m2, the doses to be given to the patients will be calculated according to BSA = 2.2 m2. No ideal body weight should be used for the calculation of BSA.

The drug is commercially available. At the discretion of the principle investigator it is possible to administer modest pre and post chemotherapy hydration, the same principle applies with regard to the preventive anti-emetic treatment to be carried out at the same time as the therapy and, if needed, at home.

The working out of the dosage of the drug to be administered must be done at the beginning of the treatment taking the body surface into account which in turn has to be worked out with respect to patient's weight and height.

At the end of the entire protocol program tumor assessment will be performed every 3 months, during follow up visit for the first two years, then from third to fifth year and until evidence of relapse or death. After relapse, follow up visit will continue until patient's death in order to collect survival data.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to a complete cytoreductive surgery and subsequent HIPEC for PMP
* Histological diagnosis of pseudomyxoma peritonei (PMP)
* Assessment of KRAS mutation positivity on surgical sample
* Age >= 18 years and <76 years
* Performance Status (ECOG <2)
* Adequate organ function including the following:
* Adequate bone marrow reserve: WBC count >3.0x109/L, absolute neutrophyl count >1.5x109/L, platelet count >100x109/L, and hemoglobin >10 g/dL
* Hepatic: bilirubin < 1.5 times the ULN, alkaline phosphatase, aspartate transaminase, and alanine transaminase < 2.5 xULN
* Renal: Creatinine clearance >50 mL/min or serum creatinine 1.5 x UNL
* Patients compliance and geographic proximity that allows for adequate follow-up
* Patients must sign an informed consent document (ICD)
* Male and female patients with reproductive potential must use an approved contraceptive method.

Exclusion Criteria:

* Previous systemic chemotherapy and/or biological therapy
* Administration of other experimental drugs during the study
* Pregnancy and breast-feeding
* Serious or uncontrolled medical pathologies or active infections that would jeopardize the possibility of receiving the investigated treatment
* Disorders that could influence the absorption of capecitabine (e.g. malabsorption), intestinal occlusion, Crohn's disease or ulcerative colitis
* Psychiatric disorders, neurologic disease or other conditions that would make it impossible to comply with the protocol procedures.
* Positive anamnesis with regard to other neoplastic diseases except for the ones that have been cured for more than 5 years

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Progression free survival is time between treatment start date and first date of recurrence or death, whichever occurs first.
  To evaluate the efficacy of postoperative capecitabine in terms of progression free survival (PFS) after CRS and HIPEC in patients with KRAS mutated PMP with extensive peritoneal disease

SECONDARY OUTCOMES:
OS | Overall survival (OS) is time between the date of chemotherapy start and the date of death. For subjects without documentation of death, OS will be censored on the last date the subject was known to be alive
  To assess the efficacy of adjuvant capecitabine treatment in terms of overall survival (OS)
DSS | Disease Specific Survival (DSS) is time between the date of chemotherapy start and the date of death caused by cancer. Deaths from other causes are not "events".
  To assess the efficacy of adjuvant capecitabine treatment in terms of isease specific survival (DSS)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Di Bartolomeo, MD, Principal Investigator — IRCCS Istituto Nazionale Tumori MIlano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, MI, Italy